CLINICAL TRIAL: NCT01533974
Title: Acceptance & Commitment Therapy for Smoking Cessation (Aka PATH Study - Partnering to Achieve Tobacco-free Health)
Brief Title: PATH Partnering to Achieve Tobacco-free Health
Acronym: PATH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IR7441
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Acceptance and Commitment Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT (Experimental): We will use a five-session (90 minutes per session) group-delivered adaptation of Dr. Bricker's ACT treatment program.
  Interventions: Other: Acceptance & Commitment Therapy (ACT)
- CBT (Active Comparator)
  Interventions: Other: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Other: Acceptance & Commitment Therapy (ACT) — We will use a five-session (90 minutes per session) group-delivered adaptation of Dr. Bricker's ACT treatment program.
  Arms: ACT
Other: Cognitive Behavioral Therapy (CBT) — The control condition will be the current group-delivered CBT smoking cessation program at GH.
  Arms: CBT

SUMMARY:
The overall aim of this 5-year project is to capitalize on the strong theoretical and promising empirical evidence for Acceptance & Commitment Therapy (ACT) as an intervention for smoking cessation by comparing the effectiveness of ACT against standard cognitive behavioral therapy (CBT) counseling when both are offered with nicotine replacement therapy (NRT) and delivered within a real world healthcare setting.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 and older;
2. smoke at least 10 cigarettes per day for every day in the past month;
3. want to quit smoking in the next 30 days;
4. are able to speak and read in English;
5. are a GH member enrolled living in the greater Seattle area;
6. are not currently participating in other smoking cessation interventions;
7. not currently using other nicotine products (e.g., smokeless tobacco)
8. are willing to attend five 90-minute group intervention sessions and to receive NRT over the next 3 months;
9. have no medical contraindications for NRT use (i.e., pregnant, breastfeeding, recent heart attack, or skin allergy preventing use of the patch, as assessed using the standard GH contraindication screening for NRT patch);
10. no household member currently enrolled in the study

Exclusion Criteria:

1. fails to meet the eligibility criteria above;
2. has a significant cognitive or physical impairment (e.g., dementia, deafness) that would preclude full participation in the counseling sessions. This will be assessed both by self-report and by in-person assessment at the baseline enrollment appointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2011-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700

RESULTS

PARTICIPANT FLOW:
Groups:
- Acceptance and Commitment Therapy (ACT): We will use a five-session (90 minutes per session) group-delivered adaptation of Dr. Bricker's ACT treatment program.
  Acceptance & Commitment Therapy (ACT): We will use a five-session (90 minutes per session) group-delivered adaptation of Dr. Bricker's ACT treatment program.
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy (ACT) | Cognitive Behavioral Therapy (CBT)
Started | 224 | 226
Completed | 173 | 176
Not Completed | 51 | 50

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy (ACT) | Cognitive Behavioral Therapy (CBT) | Total
Number analyzed (Participants) | 224 | 226 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (12.0) | 50.8 (12.2) | 51.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 119 | 237
  Male | 106 | 107 | 213

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Stopped Smoking by 12 Month Post Treatment
Description: 30 day point prevalence abstinence at 12 months. Missing = smoking and self report.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Acceptance and Commitment Therapy (ACT) | Cognitive Behavioral Therapy (CBT)
Number analyzed (Participants) | 224 | 226
participants | 31 | 41

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Acceptance and Commitment Therapy (ACT) | Cognitive Behavioral Therapy (CBT)
Serious Adverse Events (participants affected / at risk) | 0/224 | 0/226
Other Adverse Events (participants affected / at risk) | 17/224 | 5/226
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acceptance and Commitment Therapy (ACT) (N=224) | Cognitive Behavioral Therapy (CBT) (N=226)
Disturbed Sleep (General disorders) | 7 (7) | 1 (1) — Vivid, strange, weird dreams; common side effect of NRT
Skin irritation (General disorders) | 3 (3) | 1 (1) — Burning, itching, rash at patch site; common side effect of NRT.
Muscle Ache (General disorders) | 1 (1) | 1 (1) — Muscle ache and soreness at patch site; common side effect of NRT patch.
Stomach and digestive issues (General disorders) | 3 (3) | 1 (1) — Indigestion, nausea, and upset stomach; common side effect of NRT patch.
Dry mouth (General disorders) | 1 (1) | 0 (0) — Dry mouth; common side effect of NRT patch.
Headache (General disorders) | 1 (1) | 0 (0) — Headache off and on for past week; probably related
MRSA infection (General disorders) | 0 (0) | 1 (1) — Participant was treated for a MRSA infection; not related.
Anxiety (General disorders) | 1 (1) | 0 (0) — Anxiety and difficulty concentrating when first using the patch; common side effect of patch

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No